CLINICAL TRIAL: NCT00772096
Title: Septic Encephalopathy and Late Cognitive Dysfunction in Patients With Sepsis - the Role of Inflammation
Brief Title: Septic Encephalopathy and Late Cognitive Dysfunction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: EK 151/08
Record Dates: First submitted 2008-10-14; First posted 2008-10-15 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Sepsis; Severe Sepsis
MeSH Terms: conditions — Sepsis | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Verum (Experimental)
  Interventions: Drug: n-3 fatty acids
- No treatment (No Intervention)

INTERVENTIONS:
Drug: n-3 fatty acids
  Arms: Verum

SUMMARY:
Delirium and long-term cognitive dysfunction are important problems in intensive care patients. Patients with sepsis are at a high risk of developing delirium (septic encephalopathy), which may be an important risk factor for the development of long-term cognitive dysfunction.

Working hypotheses: 1. Septic encephalopathy and cognitive dysfunction are caused by an unspecific reaction of the brain to an intense inflammatory stimulus. 2. It is possible to therapeutically influence the inflammatory response and its effects on the brain.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to an intensive care unit for treatment of sepsis, severe sepsis or septic shock
* Age 18 or older

Exclusion Criteria:

* Primary infection of the CNS
* History of cerebrovascular disease
* History of any neoplasia involving the CNS
* History of long-term psychiatric medication
* History of allergy to fish- or egg-protein
* Severe coagulation abnormalities
* Clinical signs of altered coagulation, active bleeding
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luzius A Steiner, MD, PhD, Principal Investigator — Department of Anaesthesia, University Hospital Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Basel, Switzerland

REFERENCES:
- [Derived] Burkhart CS, Dell-Kuster S, Siegemund M, Pargger H, Marsch S, Strebel SP, Steiner LA. Effect of n-3 fatty acids on markers of brain injury and incidence of sepsis-associated delirium in septic patients. Acta Anaesthesiol Scand. 2014 Jul;58(6):689-700. doi: 10.1111/aas.12313. Epub 2014 Mar 24. PMID 24660837